CLINICAL TRIAL: NCT00369928
Title: A Multicenter, Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of 2 Oral Doses, 25 mg Twice Daily and 100 mg Twice Daily, of PG-760564 in Adult Patients With RA Receiving Methotrexate
Brief Title: Evaluation of 2 Oral Doses of PG-760564 in Rheumatoid Arthritis (RA) Patients Receiving Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Muhammad Rehman, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006012
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Results first posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, oral dose, BID
  Interventions: Drug: Placebo dose
- 25 mg PG-760564 (Experimental): 25 mg BID, of oral PG-760564
  Interventions: Drug: PG-760564
- 100 mg PG-760564 (Experimental): 100 mg BID, of oral PG-760564
  Interventions: Drug: PG-760564

INTERVENTIONS:
Drug: PG-760564 — 100 mg BID, of oral PG-760564
  Arms: 100 mg PG-760564
Drug: Placebo dose — placebo, BID, oral for 12 weeks
  Arms: Placebo
Drug: PG-760564 — 25 mg BID, of oral PG-760564
  Arms: 25 mg PG-760564

SUMMARY:
This will be a 12-week, double-blind, randomized, placebo-controlled, parallel group, multicenter study to evaluate the safety, efficacy, and PK of oral administration of PG-760564 in adult patients with active RA receiving treatment with MTX. Two oral doses of PG-760564 will be evaluated: 25 mg BID and 100 mg BID. The study will consist of a screening visit followed by a washout period for all disease modifying antirheumatic drugs (DMARDs) and anti-cytokine therapies except MTX. After the washout period, patients determined to be eligible will be randomized to receive either 25 mg BID or 100 mg BID of oral PG-760564, or placebo for 12 weeks. There will be 6 treatment visits and a follow-up visit 4 weeks after the last treatment visit. The primary efficacy endpoint will be the proportion of patients meeting the ACR 20 response criteria after 12 weeks of treatment.

DETAILED DESCRIPTION:
The study will be conducted in North America and Europe at approximately 50 to 60 sites. Approximately 270 patients will be randomized, of which 189 are expected to complete the study.

The study will consist of a screening visit followed by a washout period for all disease modifying antirheumatic drugs (DMARDs) and anti-cytokine therapies except MTX. The washout period will be 4 weeks for sulfasalazine, hydroxychloroquine, azathioprine, D-penicillamine, etanercept, and anakinra, 8 weeks for gold, infliximab, and adalimumab, and 12 weeks for abatacept.

After the washout period, the patients determined to be eligible will be randomized to receive either 25 mg BID or 100 mg BID of oral PG-760564, or placebo for 12 weeks. There will be 6 treatment visits (Weeks 1, 2, 4, 6, 8, and 12) and a follow-up visit 4 weeks after the last treatment visit (Week 16). Patients will not initiate new therapies until after the 4-week follow-up is completed. Liver function tests will be evaluated at every visit.

The primary efficacy endpoint will be the proportion of patients meeting the ACR 20 response criteria after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) criteria for Rheumatoid Arthritis
* Disease duration of at least 6 months
* Must be treated with Methotrexate for at least 24 weeks
* At least 6 swollen joints and 6 tender joints
* Washout required for other Disease Modifying Anti-rheumatic Drugs (DMARDs)
* Women of childbearing age and all males must use acceptable method of birth control

Exclusion Criteria:

* Tuberculosis
* Malignancies
* Abnormal electrocardiograms as described in the protocol
* Current infection or recurrent infections or immunodeficiency
* Liver diseases and abnormalities in liver function tests as described in the protocol
* Autoimmune diseases other than RA except Sjogren's syndrome secondary to RA;
* History of demyelization diseases
* Any condition that in the opinion of the investigator could be detrimental to patients enrolling in the study including clinically important changes in laboratory values and other diseases described in the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Rehman, MD, Study Director — Procter and Gamble
Locations (51):
- United States (23):
  - Research Facility, Hot Springs, Arkansas
  - Research Facility, Beverly Hills, California
  - Research Facility, Mission Viejo, California
  - Research Facility, Chiefland, Florida
  - Research Facility, Dunedin, Florida
  - Research Facility, Fort Lauderdale, Florida
  - Research Facility, Tavares, Florida
  - Research Facility, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Rome, Georgia
  - Research Facility, Meridian, Idaho
  - Research Facility, New Orleans, Louisiana
  - Research Facility, Omaha, Nebraska
  - Research Facility, Elizabeth, New Jersey
  - Research Facility, Plainview, New York
  - Research Facility, Charlotte, North Carolina
  - Research Facility, Wilmington, North Carolina
  - Research Facility, Minot, North Dakota
  - Research Facility, Duncansville, Pennsylvania
  - Research Facility, Erie, Pennsylvania
  - Research Facility, Austin, Texas
  - Research Facility, Dallas, Texas
  - Research Facility, San Antonio, Texas
- Czechia (5):
  - Research Facility, Česká Lípa
  - Research Facility, Hustopeče
  - Research Facility, Prague
  - Research Facility, Uherské Hradiště
  - Research Facility, Zlín
- Hungary (6):
  - Research Facility, Balatonfüred
  - Research Facility, Budapest
  - Research Facility, Eger
  - Research Facility, Győr
  - Research Facility, Gyula
  - Research Facility, Szolnok
- Research Facility, The Hague, Den Haag, Netherlands
- Poland (12):
  - Research Facility, Częstochowa, Częstochowa
  - Research Facility, Działdowo, Działdowo
  - Research Facility, Elblag, Elbląg
  - Research Facility, Gmina Końskie, Konskie
  - Research Facility, Krakow, Krakow
  - Research Facility, Lublin, Lublin Voivodeship
  - Research Facility, Poznan, Poznań
  - Research Facility, Sopot, Sopot
  - Research Facility, Szczecin, Szczecin
  - Research Facility, Torun, Torun
  - Research Facility, Warsaw, Warszawa
  - Research Facility, Lodz, Łódź Voivodeship
- United Kingdom (4):
  - Research Facility, Ashford, Ashford
  - Research Facility, Cambridge, Cambridge
  - Research Facility, Glasgow, Glasgow
  - Research Facility, Liverpool, Liverpool

RESULTS

PARTICIPANT FLOW:
Groups:
- 25 mg PG-760564 BID: 25 mg BID, of oral PG-760564
- 100 mg PG-760564 BID: 100 mg BID, of oral PG-760564
Period: Overall Study
Arm/Group | Placebo | 25 mg PG-760564 BID | 100 mg PG-760564 BID
Started | 85 | 85 | 86
Completed | 77 | 69 | 66
Not Completed | 8 | 16 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 25 mg PG-760564 BID | 100 mg PG-760564 BID | Total
Number analyzed (Participants) | 85 | 85 | 86 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 78 | 79 | 232
  >=65 years | 10 | 7 | 7 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 51.52 (11.04) | 50.39 (11.68) | 54.70 (9.31) | 52.21 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 66 | 195
  Male | 21 | 20 | 20 | 61
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 9 | 29
  Poland | 45 | 42 | 49 | 136
  United Kingdom | 3 | 0 | 0 | 3
  Czech Republic | 18 | 23 | 16 | 57
  Hungary | 10 | 9 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Meeting American College of Rheumatology 20 Response Criteria (ACR20) at 12weeks
Description: percent, relative to baseline, of patients meeting the American College of Rheumatology 20 response criteria (ACR20) at 12weeks
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percent meeting ACR 20
Arm/Group | Placebo | 25 mg PG-760564 BID | 100 mg PG-760564 BID
Number analyzed (Participants) | 85 | 85 | 86
percent meeting ACR 20 | 60 [48 to 72] | 56 [43 to 68] | 54 [41 to 67]
Statistical Analysis 1: Comparison: Placebo vs 25 mg PG-760564 BID; Test type: Superiority or Other; p = 0.982, Cochran-Mantel-Haenszel; Odds Ratio, log = 0.88, 80% CI 2-sided [0.56 to 1.38]
Statistical Analysis 2: Comparison: Placebo vs 100 mg PG-760564 BID; Test type: Superiority or Other; p = 0.666, Cochran-Mantel-Haenszel; Odds Ratio, log = 0.79, 80% CI 2-sided [0.50 to 1.25]

ADVERSE EVENTS:
Arm/Group | Placebo | 25 mg PG-760564 BID | 100 mg PG-760564 BID
Serious Adverse Events (participants affected / at risk) | 1/85 | 4/85 | 6/86
Other Adverse Events (participants affected / at risk) | 3/85 | 2/85 | 5/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | 25 mg PG-760564 BID (N=85) | 100 mg PG-760564 BID (N=86)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=85) | 25 mg PG-760564 BID (N=85) | 100 mg PG-760564 BID (N=86)
Alanine aminotransferase increased (Investigations) | 3 (4) | 2 (2) | 5 (5) — Alanine aminotransferase increased

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It will be the Sponsor's responsibility to convene and charter a Publications Committee consisting of representation from the Sponsor and key academic and investigational centers. The Publications Committee will be primarily responsible for the creation, review, and submission of publications and presentations relating to the major aspects of the study (design, baseline data, mortality and safety data) and ancillary analyses after the completion of the study.